CLINICAL TRIAL: NCT05821946
Title: The Effect of Web-Based Multi-source Training on the Prevention of Urinary Tract Infections in Adult Kidney Transplant Recipients on Clinical Outcomes
Brief Title: Web-Based Multi-Resource Training on the Prevention of Urinary Tract Infections in Adult Kidney Transplant Recipients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Fatma CEBECİ, Professor Doctor, Akdeniz University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: KAEK-896-2021
Record Dates: First submitted 2023-02-12; First posted 2023-04-20 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2023-10

CONDITIONS: Kidney Transplantation; Adult; Urinary Tract Infections; Prevention; Medical Informatics
Keywords: Kidney; Transplantation; Adult; Urinary Tract Infection; Prevention; Nursing; Web-Based Multi-Source Education for Patients; Medical Informatics
MeSH Terms: conditions — Urinary Tract Infections

STUDY DESIGN:
Intervention Model Description: The study is a single-center, parallel-group, single-blind, pretest, and posttest randomized controlled experimental study.
Who Masked: Participant, Outcomes Assessor
Masking Description: In the research, the participants will be blinded; the researcher cannot be blinded because he is practicing. To avoid statistical evaluator bias, statistical evaluations will be made on a data file where the intervention or control group is not explicitly stated by the researcher.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Web-Based Multi-Source Training on the Prevention of Urinary Tract İnfections (Experimental): In addition to routine training, web-based multi-source training will be provided on the prevention of urinary tract infections in adult kidney transplant recipients.
  Interventions: Other: Web-Based Multi-Source Training on the Prevention of Urinary Tract İnfections
- Control group (No Intervention): Routine training and before discharge will be directed to the organ transplant handbook on the transplant center's website.

INTERVENTIONS:
Other: Web-Based Multi-Source Training on the Prevention of Urinary Tract İnfections — Before discharge, individuals will be given a user name and password to enter the website by the researcher. The first access to the website will be made via the researcher's computer, and the website will be introduced. Individuals will be shown how to access the compatible website on Android and IOS phones and tablets by the researcher. Web-based multi-source training for individuals to prevent urinary tract infections will begin. The researcher will check the use of educational materials by individuals from the administrator's menu. To increase the effectiveness of the training, reminder, motivating, and supportive messages will be sent to the patients twice a week.
  Arms: Web-Based Multi-Source Training on the Prevention of Urinary Tract İnfections

SUMMARY:
Purpose: The study aims to examine the effect of web-based multi-source training on the prevention of urinary tract infections in adult kidney transplant recipients on clinical outcomes.

Design: The study is a single-center, parallel-group, single-blind, pretest, and posttest randomized controlled experimental study.

Methods: A total of 90 kidney transplant recipients, 45 in the control group and 45 in the intervention group will be included in the study. Kidney transplant recipients will be randomized on the day of discharge. Before discharge, the Patient Socio-Demographical/Descriptive Characteristics Form and the Discharge Readiness Scale will be applied to the control and intervention groups. Routine training and aimed at preventing urinary tract infections web-based multi-source training will be provided to the intervention group. The developed educational material was evaluated by experts in terms of literacy, reliability, and information quality. As multiple resources on the web: there will be written and visual texts of the educational material, as well as podcasts and animation videos. Web page usability will be evaluated with the System Usability Scale. Individuals will be able to benefit from each of these multiple educational resources according to their preferences. The control group will be directed to the organ transplantation handbook on the website of the routine education and organ transplant center. After discharge, the follow-ups of the intervention and control group were carried out during the first 6-month post-transplant standard follow-up process of the center (2. day; once a week for the first month; every ten days for up to 1-3 months; every three weeks for the next 3-6 months) will be performed. When patients come to their controls, the results of routine examinations (complete urinalysis, urine culture taken when necessary, hospitalization, emergency application, and other data) will be taken from the Hospital Information Management System. In addition, the recipients' opinions in the intervention group on the Web-Based Multi-Resource Training Program will also be received at the end of the 6th month. The research adhered to the Standard Protocol Items: Recommendations for Interventional Trials-SPIRIT (2013) and Consolidated Standards of Reporting Trials-CONSORT (2018) checklists.

DETAILED DESCRIPTION:
1. INTRODUCTION

   Kidney transplant (KTx) is the most common and successful treatment of all types of organ replacement. However, urinary tract infections (UTIs), commonly seen in kidney transplant recipients, negatively affect successfully performed kidney transplantation. Therefore, prevention and effective infection treatment are of great importance to optimize, maintain, and prolong the function of the graft and avoid rejection in KTx recipients. Although UTIs can occur at any time after transplantation, they are more common in the early stages of KTx. Urinary tract infections cause frequent hospital admissions and repeated hospitalizations. This situation causes frequent hospital admissions and repeated hospitalizations of patients. Post-kidney transplant UTIs with high recurrence rates burden health economics and treatment outcomes.

   Websites compatible with mobile devices, one of the methods of meeting health needs, significantly affect people's ability to manage their health and acquire long-term healthy lifestyle behaviors. It also can reduce health expenditures. However, in the literature review, there were no studies examining the effect of education and training to prevent urinary tract infections in adult KTx recipients on clinical outcomes. The aim of this study was to evaluate the effect of web-based multi-source training on clinical outcomes in adult kidney transplant recipients to prevent urinary tract infections.

   The following hypotheses will be tested.

   H1-1: The effect of web-based multi-source education to prevent UTIs in adult kidney transplant recipients on infection is significantly different than in the control group.

   H1-2: The effect of web-based multi-source education to prevent UTIs in adult kidney transplant recipients on the number of emergency visits is significantly different than in the control group.

   H1-3: The effect of web-based multi-source education to prevent UTIs in adult kidney transplant recipients on hospital readmission is significantly different than in the control group.

   H1-4: Adult kidney transplant recipients who are ready for discharge versus those who are not ready for release are significantly different in clinical outcomes.
2. METHODS

Study design

This study is a single-center, parallel-group, single-blind, pre-test and post-test randomized controlled experimental study. The research will begin after obtaining the ethics committee's approval, institutional permission, and informed consent. In the study, Standard Protocol Items: Recommendations for Interventional Trials-SPIRIT and Consolidated Standards of Reporting Trials-CONSORT checklists will be adhered to.

The sample size was calculated using the calculation formula with the known universe and the Raosoft sample size calculation online application. In a study of kidney transplant recipients, the urinary tract infection rate was 25.2%. Considering this finding, the minimum sample size was calculated as 85 with a 95% confidence interval and a 5% deviation. The patients to be sampled will be determined by stratified random sampling method (stratification criterion: Gender). When proportioned according to the layer weights, 60 male and 25 female patients will be included in the study. Considering the losses experienced during the research, 90 patients who meet the inclusion criteria will be included in the sample. Individuals included in the study will be assigned to the intervention (45) and control (45) groups.

Randomization and allocation

Randomization will be done by an independent person from the research team on https://www.randomizer.org/. According to the randomization results, a list will be created for the patients. The research participants will be shown in the CONSORT flowchart. In the study, it will be stratified by gender (male, female) to ensure homogeneity between the patients in the control and intervention groups and to control the factors affecting urinary tract infections. The study will be carried out with adult kidney transplant recipients at Akdeniz University Hospital were followed up in the Outpatient Follow-up Unit.

Data will be collected using the Patient Socio-Demographical/Descriptive Characteristics Form, Scale of Readiness to Discharge, and Post-Discharge Patient Data Form. In addition to routine training for the intervention group, the website created to prevent urinary tract infections before discharge will be introduced and training. On the other hand, the control group will be directed to the training area the organ transplant website for with the handbook without being discharged, in addition to the routine training. After discharge, follow-up of the intervention and control groups will be done with the center's standard follow-up process the first six months after transplantation (day 2; weekly for the first month; every ten days for up to 1-3 months; every three weeks for the next 3-6 months).When the patients come to their controls after discharge, the results of routine examinations (complete urinalysis, urine culture taken, when necessary, hospitalization, emergency application, and other data) will be taken from the Hospital Information Management System. At the end of the 6th month, the Opinion Form on the Web-Based Multi-Resource Education Program will be applied to kidney recipients in the intervention group.

Developing and Implementing Web-Based Multi-Source Education

Web-based multi-source educational content to prevent UTIs in adult KTx recipients was prepared using the literature. Educational content to prevent UTIs; the importance of urinary system infection in kidney transplantation, urinary system, UTIs, symptom findings, diagnosis, sampling for urine culture, adequate fluid intake, diabetes management, healthy toilet habits, genital hygiene, and other hygiene recommendations, healthy sexual intercourse and birth control measures, healthy and balanced diet, obesity prevention, urinary catheter care, physical activity, drug use recommendations. After the written training material was prepared, its readability by adult kidney transplant recipients was calculated according to the Turkish readability formula.

The literacy of the developed training material: The Appropriateness of Written Materials Evaluation Form reliability and information quality with the DISCERN (Quality Criteria for Consumer Health Information) Scale evaluated by 15 experts. The Web site to be created to prevent urinary tract infections in adult kidney transplant recipients will include written and visual educational materials, podcasts, and animation videos as multiple educational resources. Individuals can benefit from these multiple educational resources according to their preferences. Moving visual content and audio elements will be balanced in educational materials, podcasts, and animation videos prepared by the researcher. In addition to these, while the visuals are being crafted, buttons, pop-ups, shapes, and podcast audio applications will be designed by the understanding level and expectations of the target audience. A web page design and design compatible with android and IOS phones, computers, and tablets will be prepared by an expert software developer. The prepared web program is compatible with computers, tablets, and mobile devices and the website can use on every platform easily.

Interventions

Interventions will be implemented by Kiraz according to the study protocol established by Kiraz and Cebeci.

Trial organization

The coordination center is located in Antalya, Akdeniz University Prof. Dr. Tuncer KARPUZOĞLU is at the Organ Transplantation Institute. This group is responsible for the overall design and progress of the research.

Membership: FC, NK

Limitations

The research data are limited to patients in the 18-65 age group who underwent kidney transplantation and follow-up at Akdeniz University Hospital.

ELIGIBILITY:
Inclusion criteria

* 18-65 years
* Ability to speak, read and write Turkish.
* Becoming a kidney transplant recipient for the first time
* Having and using a smartphone (IOS or Android) or computer or tablet
* Having internet access

Exclusion criteria

* Willingness to leave the research at any time
* Re-operation in the follow-up process
* Hospitalization due to non-transplant problems during follow-up
* Not using the web-based application despite three reminder messages a week.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Infection status | Up to 6 months after discharge
  The urinary tract infection status of kidney transplant recipients will be evaluated by obtaining the results of routine examinations performed at standard controls after discharge from the Hospital Information Management System.
Number of applications to the emergency department | Up to 6 months after discharge
  The number of applications to the emergency department due to urinary tract infections of kidney transplant recipients will be obtained from the Hospital Information Management System.
Hospital readmission status | Up to 6 months after discharge
  Re-hospitalization status of kidney transplant recipients due to urinary tract infection will be obtained from the Hospital Information Management System.

SECONDARY OUTCOMES:
Adult kidney transplant recipients who are ready for discharge versus those who are not ready for release are significantly different in clinical outcomes. | Within 24 hours before discharge
  The Readiness for Hospital Discharge Scale/Short Form will be used to evaluate the patient's readiness for discharge. The scale consists of eight items and four dimensions, and the items in the hierarchy are assessed on a scale ranging from 0 to 10. Dimensions of the scale; the patient's situation, the patient's knowledge, the patient's coping skills, and the patient's expected support. If the score of the scale dimensions is ≥7, the patient is considered ready for discharge, and if it is <7, the patient is considered not prepared.
Views of adult kidney transplant recipients on web-based multi-source urinary tract infection prevention education | End of 6 months after discharge
  The opinions and satisfactions of adult kidney transplant recipients in the intervention group regarding the web-based multi-source training program will be evaluated with 3 open-ended questions at the end of the 6-month follow-up period after transplantation.

CONTACTS AND LOCATIONS:
Overall Officials: Fatma CEBECİ, Principal Investigator — Akdeniz University; Nihal KİRAZ, Principal Investigator — Akdeniz University
Locations (1):
- Akdeniz University, Antalya, Turkey (Türkiye)